CLINICAL TRIAL: NCT02714049
Title: Two Arm Open Label Pilot Study of Flibanserin (Addyi®) vs. Flibanserin and Sex Therapy
Brief Title: Flibanserin (Addyi®) vs. Flibanserin and Sex Therapy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Investor Initiated Grant support stopped when drug was sold.
Sponsor: San Diego Sexual Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDSM-2015-03
Record Dates: First submitted 2016-03-11; First posted 2016-03-21 (Estimated); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Hypoactive Sexual Desire Disorder
Keywords: hypoactive sexual desire disorder; Addyi; flibanserin; low sexual desire; HSDD
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — Psychotherapy; flibanserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- flibanserin (Experimental): Subjects meeting inclusion/exclusion criteria who respond to flibanserin will have a total of 20 weeks of open label drug
  Interventions: Drug: flibanserin
- flibanserin and sex therapy (Experimental): Subjects meeting inclusion/exclusion criteria who respond to flibanserin will have a total of 20 weeks of open label drug as well as 9 sex therapy visits
  Interventions: Behavioral: sex therapy; Drug: flibanserin

INTERVENTIONS:
Behavioral: sex therapy — 60 minutes each time, in person or on the telephone
  Other Names: psychotherapy
  Arms: flibanserin and sex therapy
Drug: flibanserin — FDA approved medication for treatment of hypoactive sexual desire disorder in premenopausal women
  Other Names: Addyi

SUMMARY:
Unblinded study of flibanserin for 8 weeks with responders randomized 1:1 to receive study medication alone vs. study medication and sex therapy for 12 additional weeks.

DETAILED DESCRIPTION:
This is an unblinded study to be conducted at a single research center, San Diego Sexual Medicine. Subjects meeting inclusion and exclusion criteria will receive flibanserin for an 8-week run-in period to differentiate between responders and non-responders. Responders will be determined by a score of 1-3 on the Patient Global Impression of Improvement (PGI-I) at 8 weeks from baseline, and will be randomized 1:1 to receive study medication alone vs. study medication and sex therapy for an additional 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing and able to provide written informed consent and HIPAA authorization before any study procedures are conducted;
2. Subject is female;
3. Subject is ≥18 years old;
4. Subject has biologic-based HSDD as her primary sexual complaint;
5. Subject scores <26 on FSFI and <4.8 on desire domain of FSFI at screening;
6. Subject scores >18 on FSDS-DAO;
7. Subject answers yes to questions 1-4 on the DSDS screener;
8. Subject is willing to use effective contraception during the study if pre-menopausal (oral contraceptives, barrier method, long acting reversible contraceptive, surgical sterilization);
9. Subject agrees to comply with the study procedures and visits.

Exclusion Criteria:

1. Subject has sexual pain;
2. Subject does not have generalized, acquired HSDD;
3. Subject has used flibanserin in the last 6 months;
4. Subject has history of alcohol or drug abuse;
5. Subject uses tobacco in any form;
6. Subject is currently using androgen therapy and unwilling to washout;
7. Subject is pregnant, nursing, or planning to become pregnant over the next 6 months;
8. Subject is taking a moderate or strong cytochrome P450 3A4 (CYP3A4) inhibitor;
9. Subject is taking a CYP3A4 inducer;
10. P-glycoprotein substrate;
11. Subject has a history of liver impairment;
12. Subject has any chronic medical condition or psychologic disorder that the Principal Investigator feels makes her ineligible for the study;
13. Subject has any condition or exhibits behavior that indicates to the Principal Investigator that the Subject is unlikely to be compliant with study procedures and visits.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Desire domain of the Female Sexual Function Index (FSFI) | at weeks 8 and 20
  The primary objective of this study is to determine whether efficacy of flibanserin as determined by changes in the desire domain of the Female Sexual Function Index (FSFI) in women who respond to the study medication is greater when sex therapy is performed concomitant with the use of the medication.

SECONDARY OUTCOMES:
Female Sexual Distress Scale (FSDS-DAO) | at weeks 8 and 20
  One secondary endpoint is to determine whether efficacy of flibanserin as determined by changes from baseline in the Female Sexual Distress Scale (FSDS-DAO) in women who respond to the study medication.
Total score of the Female Sexual Function Index (FSFI) | at weeks 8 and 20
  One secondary endpoint is to determine whether efficacy of flibanserin as determined by changes from baseline in the total FSFI score respectively in women who respond to the study medication.

OTHER OUTCOMES:
Patient Global Impression of Improvement (PGI-I) | at weeks 8 and 20
  The last goal is to identify those women with primary biologic based HSDD who respond to flibanserin and determine whether or not they feel concomitant sex therapy might be more beneficial.

CONTACTS AND LOCATIONS:
Overall Officials: Irwin Goldstein, MD, Principal Investigator — San Diego Sexual Medicine
Locations (1):
- San Diego Sexual Medicine, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical trials at San Diego Sexual Medicine — https://www.sandiegosexualmedicine.com/clinical-trials